CLINICAL TRIAL: NCT06925022
Title: Educational Programs Based on Healthy Habits to Improve Quality of Life and Psychosocial Profile in Women With Neurodegenerative Diseases: The ADVICE Protocol Study
Brief Title: Educational Programs Based on Healthy Habits to Improve Quality of Life and Psychosocial Profile in Women With Neurodegenerative Diseases: The ADVICE Protocol Study (Phase 1)
Acronym: ADVICE Phase 1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Catholic University of Murcia (Other); Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Jacobo Á. Rubio-Arias, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UALBIO2021/026; PID2021-123447OA-I00 (Other Grant/Funding Number: MCIN/AEI /10.13039/501100011033 and by FEDER, UE.)
Record Dates: First submitted 2025-02-20; First posted 2025-04-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting
Keywords: Lifestyle Interventions; Menstrual Cycle; Multiple Sclerosis; Exercise; Cognitive-behavioral intervention; Physical Activity, Psychosocial Well-being; Nutrition intervention
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Women with and without multiple sclerosis will participate in a strength training session during three phases of the menstrual cycle: early follicular phase, late follicular phase, and mid-luteal phase. Before and after each session, various measurements will be taken to assess physiological and performance responses.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this study, double blinding will be implemented to reduce bias in data collection. On one hand, the participants will not know which phase of the menstrual cycle they are in at the time of evaluation. For this purpose, the scheduling of measurements will be based on prior records. On the other hand, the researchers will also be unaware of the menstrual cycle phase. The assignment of phases and groups will be managed by an independent study coordinator who will not participate in direct evaluations. Additionally, the data will be coded to ensure that evaluators cannot identify the study variables during the measurement process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women with MS (Experimental): This arm will comprise women diagnosed with relapsing-remitting Multiple Sclerosis (RRMS) according to the McDonald criteria.
  Interventions: Other: Strength training session during Early Follicular Phase; Other: Strength Training Protocol during Late Follicular Phase; Other: Strength Training during Mid-Luteal Phase
- Women without Multiple Sclerosis (Other): This arm will comprise women without Multiple Sclerosis, matched with the MS group based on age, lifestyle habits, and geographic location.
  Interventions: Other: Strength training session during Early Follicular Phase; Other: Strength Training Protocol during Late Follicular Phase; Other: Strength Training during Mid-Luteal Phase

INTERVENTIONS:
Other: Strength training session during Early Follicular Phase — The strength training sessions follow guidelines and recent meta-analyses to optimize long-term outcomes. Participants will complete a standardized warm-up protocol consisting of 5 minutes on a stationary bike, lower limb mobility exercises, and 5 repetitions at 40% of their 1-RM on each machine before each strength training session. Subsequently, they will perform four exercises for the lower limbs, including bilateral leg press, unilateral leg extension, unilateral hip extension, and plantar flexion, using conventional weight machines (. Session intensity will be set at 70-75% of 1-RM, with a volume of 4 sets of 10 repetitions, leaving 1-2 reps in reserve (RIR), and with 120 seconds of rest between sets.
  This phase occurs at the beginning of the menstrual cycle (days 2-5 after the onset of menstruation).
Other: Strength Training Protocol during Late Follicular Phase — The strength training sessions follow guidelines and recent meta-analyses to optimize long-term outcomes. Participants will complete a standardized warm-up protocol consisting of 5 minutes on a stationary bike, lower limb mobility exercises, and 5 repetitions at 40% of their 1-RM on each machine before each strength training session. Subsequently, they will perform four exercises for the lower limbs, including bilateral leg press, unilateral leg extension, unilateral hip extension, and plantar flexion, using conventional weight machines (. Session intensity will be set at 70-75% of 1-RM, with a volume of 4 sets of 10 repetitions, leaving 1-2 reps in reserve (RIR), and with 120 seconds of rest between sets. This phase occurs approximately between days 11-13 of the menstrual cycle.
Other: Strength Training during Mid-Luteal Phase — The strength training sessions follow guidelines and recent meta-analyses to optimize long-term outcomes. Participants will complete a standardized warm-up protocol consisting of 5 minutes on a stationary bike, lower limb mobility exercises, and 5 repetitions at 40% of their 1-RM on each machine before each strength training session. Subsequently, they will perform four exercises for the lower limbs, including bilateral leg press, unilateral leg extension, unilateral hip extension, and plantar flexion, using conventional weight machines (. Session intensity will be set at 70-75% of 1-RM, with a volume of 4 sets of 10 repetitions, leaving 1-2 reps in reserve (RIR), and with 120 seconds of rest between sets. This phase occurs around days 19-28 of the menstrual cycle, following ovulation.

SUMMARY:
This phase of the project aims to analyze the interaction between physical exercise and the phases of the menstrual cycle, evaluating its impact on fatigue, functional capacity, and exercise perception in women with and without Multiple Sclerosis. To achieve this, a controlled, single-blind, prospective, 2x3 crossover, randomized clinical trial will be conducted, involving women with Multiple Sclerosis (MS), matched by age, lifestyle habits (smoking, physical activity), and geographic location with a group of women without MS. This study, aligned with previous findings, seeks to deepen the understanding of the role of exercise in managing Multiple Sclerosis symptoms and to promote greater adherence to personalized physical activity programs adapted to the phases of the menstrual cycle.

ELIGIBILITY:
Inclusion criteria include:

* Women of reproductive age (18-50 years) with MS will be included, with the upper age limit adjusted to reflect the reproductive phase;.
* No iron-deficiency anemia.
* Stable disease phase.
* Independent walking ability for over 10 meters.

Women will be recruited first and later matched with men based on age, EDSS, and lifestyle habits (physical activity, smoking, and alcohol consumption).

Exclusion criteria will include participants with MS who:

* Score <1 or >6 on the EDSS.
* Report a relapse within 12 months before the study begins.
* Have taken corticosteroid treatment within the last 2 months.
* Have participated in a structured training program in the previous 6 months.

Once all women with MS are recruited, male participants will be recruited following a 1:1 matching methodology based on age, geographic region, and lifestyle habits.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with Physical Activity | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Satisfaction with Physical Activity will be measured using an 8-item scale. Items are rated on a 5-point Likert scale ranging from 1 (Totally disagree) to 5 (Totally agree). Total scores range from 8 to 40, with higher scores indicating greater satisfaction with physical activity.
Modified Fatigue Impact Scale (MFIS) | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Fatigue perception will be measured using the MFIS. This scale is a 21-item multidimensional questionnaire that evaluates the physical, cognitive, and psychosocial effects of fatigue on a five-point ordinal scale (with a maximum total score of 84).
Modified Fatigue Impact Scale (MFIS) | Post-intervention (24 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Fatigue perception will be measured using the MFIS. This scale is a 21-item multidimensional questionnaire that evaluates the physical, cognitive, and psychosocial effects of fatigue on a five-point ordinal scale (with a maximum total score of 84).
Modified Fatigue Impact Scale (MFIS) | Post-intervention (48 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Fatigue perception will be measured using the MFIS. This scale is a 21-item multidimensional questionnaire that evaluates the physical, cognitive, and psychosocial effects of fatigue on a five-point ordinal scale (with a maximum total score of 84).
Modified Fatigue Impact Scale (MFIS) | Post-intervention (72 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Fatigue perception will be measured using the MFIS. This scale is a 21-item multidimensional questionnaire that evaluates the physical, cognitive, and psychosocial effects of fatigue on a five-point ordinal scale (with a maximum total score of 84).
Visual Analogue Scale (VAS-F): Fatigue subscale | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Fatigue (VAS-F) assesses subjective perceptions of fatigue on a scale from 0 to 10, where 0 indicates no fatigue at all and 10 indicates extreme fatigue. Higher scores reflect greater perceived fatigue.
Visual Analogue Scale (VAS-F): Fatigue subscale | Post-intervention (24 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Fatigue (VAS-F) assesses subjective perceptions of fatigue on a scale from 0 to 10, where 0 indicates no fatigue at all and 10 indicates extreme fatigue. Higher scores reflect greater perceived fatigue.
Visual Analogue Scale (VAS-F): Fatigue subscale | Post-intervention (48 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Fatigue (VAS-F) assesses subjective perceptions of fatigue on a scale from 0 to 10, where 0 indicates no fatigue at all and 10 indicates extreme fatigue. Higher scores reflect greater perceived fatigue.
Visual Analogue Scale (VAS-F): Fatigue subscale | Post-intervention (72 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Fatigue (VAS-F) assesses subjective perceptions of fatigue on a scale from 0 to 10, where 0 indicates no fatigue at all and 10 indicates extreme fatigue. Higher scores reflect greater perceived fatigue.
Visual Analogue Scale (VAS-E): Energy subscale | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Energy (VAS-E) assesses subjective perceptions of Energy on a scale from 0 to 10, where 0 indicates no energy at all and 10 indicates maximum energy. Higher scores reflect greater perceived energy.
Visual Analogue Scale (VAS-E): Energy subscale | Post-intervention (24 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Energy (VAS-E) assesses subjective perceptions of Energy on a scale from 0 to 10, where 0 indicates no energy at all and 10 indicates maximum energy. Higher scores reflect greater perceived energy.
Visual Analogue Scale (VAS-E): Energy subscale | Post-intervention (48 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Energy (VAS-E) assesses subjective perceptions of Energy on a scale from 0 to 10, where 0 indicates no energy at all and 10 indicates maximum energy. Higher scores reflect greater perceived energy.
Visual Analogue Scale (VAS-E): Energy subscale | Post-intervention (72 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Energy (VAS-E) assesses subjective perceptions of Energy on a scale from 0 to 10, where 0 indicates no energy at all and 10 indicates maximum energy. Higher scores reflect greater perceived energy.
Visual Analogue Scale (VAS-P): Pain subscale | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Pain (VAS-P) assesses subjective perceptions of pain on a scale from 0 to 10, where 0 indicates no pain at all and 10 indicates worst possible pain. Higher scores reflect greater perceived pain.
Visual Analogue Scale (VAS-P): Pain subscale | Post-intervention (24 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Pain (VAS-P) assesses subjective perceptions of pain on a scale from 0 to 10, where 0 indicates no pain at all and 10 indicates worst possible pain. Higher scores reflect greater perceived pain.
Visual Analogue Scale (VAS-P): Pain subscale | Post-intervention (48 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Pain (VAS-P) assesses subjective perceptions of pain on a scale from 0 to 10, where 0 indicates no pain at all and 10 indicates worst possible pain. Higher scores reflect greater perceived pain.
Visual Analogue Scale (VAS-P): Pain subscale | Post-intervention (72 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Visual Analogue Scale for Pain (VAS-P) assesses subjective perceptions of pain on a scale from 0 to 10, where 0 indicates no pain at all and 10 indicates worst possible pain. Higher scores reflect greater perceived pain.

SECONDARY OUTCOMES:
Muscle oxygen saturation (SMO2) | During intervention in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Muscle oxygen saturation (SMO2) will be measured in both the right and left lateral quadriceps using the Moxy 3-Sensor Bundle (Fortiori Design LLC, Hutchinson, USA), allowing for the calculation of mean SMO2 across the entire training session.
Capillary lactate concentration | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Lactate concentration will be assessed with a lactate analyzer (Lactate Scout system, RedMed, Warsaw, Poland) using fingertip capillary blood samples.
Capillary lactate concentration | During intervention in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Lactate concentration will be assessed with a lactate analyzer (Lactate Scout system, RedMed, Warsaw, Poland) using fingertip capillary blood samples.
Heart rate variability | During intervention in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  HRV measurements will be taken using a Polar H10 heart rate sensor (Kempele, Finland), which will record heartbeats during sleep. The HRV variables will be analyzed using Kubios HRV software (version 3.0). The Poincaré plot and time and frequency domains will be analyzed.
Thyroid Stimulating Hormone (TSH) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Serum TSH will be analyzed to assess thyroid function and hormonal regulation. Unit of measure: μIU/mL
Interferon-gamma (IFN-γ) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Serum levels of IFN-γ will be analyzed to assess pro-inflammatory immune response activity. Unit of measure: pg/mL
Interferon-gamma (IFN-γ) | Post-intervention (30 min after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Serum levels of IFN-γ will be analyzed to assess pro-inflammatory immune response activity. Unit of measure: pg/mL
Cognitive Function | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Brain-Derived Neurotrophic Factor (BDNF) is a protein involved in neuroplasticity, cognitive function, and neuronal survival, serving as a blood biomarker for brain health and adaptability
Cognitive Function | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Brain-Derived Neurotrophic Factor (BDNF) is a protein involved in neuroplasticity, cognitive function, and neuronal survival, serving as a blood biomarker for brain health and adaptability
Neurofilament Light Chain (NFL) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Neurofilament light chain (NFL) is one of the most relevant biomarkers in multiple sclerosis (MS). The Simoa detection technique (ultrasensitive single-molecule array) allows its analysis in serum, providing both the total value and the Z-Score, enabling precise assessment of axonal damage and disease progression.
Neurofilament Light Chain (NFL) | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Neurofilament light chain (NFL) is one of the most relevant biomarkers in multiple sclerosis (MS). The Simoa detection technique (ultrasensitive single-molecule array) allows its analysis in serum, providing both the total value and the Z-Score, enabling precise assessment of axonal damage and disease progression.
Physical Self-Perception (PSP) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Physical self-perception will be evaluated using the Physical Self-Perception Profile (PSPP), which includes six subscales: sports competence, physical condition, body attractiveness, physical strength, general physical self-perception, and overall self-perception. Each item is rated on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate more positive self-perceptions in the respective domains.
Pain Catastrophizing Scale (PCS) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS), which includes 13 items divided into three subscales: rumination, magnification, and helplessness. Participants respond using a 5-point Likert scale, ranging from 0 (not at all) to 4 (all the time). Higher scores indicate greater levels of pain catastrophizing. The total PCS score ranges from 0 to 52.
Quality of Life questionnaire (MSQOL-54) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Quality of life will be assessed using the Multiple Sclerosis Quality of Life-54 (MSQOL-54), a multidimensional health-related quality of life instrument developed specifically for individuals with multiple sclerosis. It includes 14 subscales:
  Physical Function (10-100) Role Limitations-Physical (0-100) Role Limitations-Emotional (0-100) Pain (0-100) Emotional Well-being (0-100) Energy (0-100) Health Perceptions (0-100) Social Function (0-100) Cognitive Function (0-100) Health Distress (0-100) Sexual Function (0-100) Sexual Satisfaction (0-100) Change in Health (0-100) Overall Quality of Life (0-100)
  The questionnaire also yields two composite summary scores:
  Physical Health Composite Score Mental Health Composite Score Each subscale score and composite score ranges from 0 to 100, with higher scores indicating better quality of life.
State-Trait Anxiety (STAI) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  State and Trait Anxiety will be assessed using the State-Trait Anxiety Inventory (STAI), a widely used instrument developed by Spielberger et al. It consists of two subscales:
  State Anxiety (STAI-S) - evaluates how respondents feel "right now, at this moment"
  Trait Anxiety (STAI-T) - evaluates how respondents "generally feel"
  Each subscale contains 20 items, rated on a 4-point Likert scale:
  For STAI-S: from 1 (Not at all) to 4 (Very much so)
  For STAI-T: from 1 (Almost never) to 4 (Almost always)
  Scores for each subscale range from 20 to 80, with higher scores indicating greater anxiety levels.
Rate of force development | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Participants will sit in a chair with both legs flexed at a 90-degree angle, and the tested ankle securely attached to a customized device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway). They will perform three maximum contractions, each lasting 2 seconds, with 3 minutes of rest in between. The RFD will be analyzed. Testing will begin with the right leg, and the repetition with the highest recorded value for each leg will be used in the analysis
Rate of force development | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Participants will sit in a chair with both legs flexed at a 90-degree angle, and the tested ankle securely attached to a customized device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway). They will perform three maximum contractions, each lasting 2 seconds, with 3 minutes of rest in between. The RFD will be analyzed. Testing will begin with the right leg, and the repetition with the highest recorded value for each leg will be used in the analysis
Maximum Voluntary Isometric Contraction | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Participants will sit in a chair with both legs flexed at a 90-degree angle, and the tested ankle securely attached to a customized device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway).Participants will perform three 5-second MVIC, with 3 minutes of rest in between. Testing will always begin with the right leg, and the contraction with the highest recorded MVIC value will be used in the analysis Time Frame: Before the first training session
Maximum Voluntary Isometric Contraction | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Participants will sit in a chair with both legs flexed at a 90-degree angle, and the tested ankle securely attached to a customized device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway).Participants will perform three 5-second MVIC, with 3 minutes of rest in between. Testing will always begin with the right leg, and the contraction with the highest recorded MVIC value will be used in the analysis Time Frame: Before the first training session
Maximal neural drive | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  To measure neural drive, the electromyographic activity (sEMG) of the right leg's vastus lateralis will be recorded during the MVIC (Delsys Trigno, Delsys Inc., Boston, MA) with skin prepared and electrode positioning following SENIAM guidelines. EMG peak will be analyzed. The EMG peak during MVIC will represent the maximum neural drive
Maximal neural drive | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  To measure neural drive, the electromyographic activity (sEMG) of the right leg's vastus lateralis will be recorded during the MVIC (Delsys Trigno, Delsys Inc., Boston, MA) with skin prepared and electrode positioning following SENIAM guidelines. EMG peak will be analyzed. The EMG peak during MVIC will represent the maximum neural drive
Central activation ratio | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Two bipolar electrodes (10×15 cm) will be placed on the right quadriceps, with electrical stimulation controlled by Signal 6.0 software (CED, Cambridge, England) at 100 Hz frequency, 50 pulses, 0.009 s pulse duration, and 0.01 s interval, set to 40-50% of MVIC. Central activation ratio (CAR) will be assessed through a sequence of one supramaximal twitch, a 100 Hz tetanic train, an MVIC with superimposed tetanic train, followed by a potentiated tetanic train and a potentiated supramaximal twitch. This sequence will be repeated twice with 2-minute rests, and twitch-to-tetanus ratio, MVIC peak, and maximum force values will be calculated for CAR. The CAR will be calculated using the following formula: "CAR= " "Force during MVIC" /"Force during MVIC + supramaximal stimulation"
Central activation ratio | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Two bipolar electrodes (10×15 cm) will be placed on the right quadriceps, with electrical stimulation controlled by Signal 6.0 software (CED, Cambridge, England) at 100 Hz frequency, 50 pulses, 0.009 s pulse duration, and 0.01 s interval, set to 40-50% of MVIC. Central activation ratio (CAR) will be assessed through a sequence of one supramaximal twitch, a 100 Hz tetanic train, an MVIC with superimposed tetanic train, followed by a potentiated tetanic train and a potentiated supramaximal twitch. This sequence will be repeated twice with 2-minute rests, and twitch-to-tetanus ratio, MVIC peak, and maximum force values will be calculated for CAR. The CAR will be calculated using the following formula: "CAR= " "Force during MVIC" /"Force during MVIC + supramaximal stimulation"
Upper Limb Maximum Strength | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Isometric grip strength will be measured with an electronic dynamometer (K-Force Grip, Kinvent, Montpellier, France) as participants stand with elbows extended. Each hand will perform 3 trials, with 30 seconds rest between attempts
Upper Limb Maximum Strength | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Isometric grip strength will be measured with an electronic dynamometer (K-Force Grip, Kinvent, Montpellier, France) as participants stand with elbows extended. Each hand will perform 3 trials, with 30 seconds rest between attempts
Spasticity | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Pendulum Test is used to assess the level of spasticity by evaluating the resistance to passive movement in the affected limb. The test involves moving the limb in a pendulum-like motion and observing the fluidity of the movement, with increased resistance indicating higher spasticity levels
Spasticity | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The Pendulum Test is used to assess the level of spasticity by evaluating the resistance to passive movement in the affected limb. The test involves moving the limb in a pendulum-like motion and observing the fluidity of the movement, with increased resistance indicating higher spasticity levels
Intrinsic muscle characteristics: Tone (F) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Tone assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia). Definition: Oscillation frequency [Hz] that characterizes the intrinsic tension of biological soft tissues at the cellular level.
Intrinsic muscle characteristics: Tone (F) | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Tone assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia). Definition: Oscillation frequency [Hz] that characterizes the intrinsic tension of biological soft tissues at the cellular level.
Gait speed | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Gait speed will be determined with the 10-meter walk test using two photocells (Ergotest Technology AS, Langesund, Norway) at 5 and 10 meters; participants will complete two maximum-speed trials, with the slower time recorded
Gait speed | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Gait speed will be determined with the 10-meter walk test using two photocells (Ergotest Technology AS, Langesund, Norway) at 5 and 10 meters; participants will complete two maximum-speed trials, with the slower time recorded
Static balance with eyes open | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Balance is measured with static trials on a force platform (Ergotest Technology AS, Langesund, Norway), where participants stand barefoot with arms at their sides for two 30-second trials each
Static balance with eyes open | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Balance is measured with static trials on a force platform (Ergotest Technology AS, Langesund, Norway), where participants stand barefoot with arms at their sides for two 30-second trials each
Static balance with eyes closed | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Balance is measured with static trials on a force platform (Ergotest Technology AS, Langesund, Norway), where participants stand barefoot with arms at their sides for two 30-second trials each
Static balance with eyes closed | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Balance is measured with static trials on a force platform (Ergotest Technology AS, Langesund, Norway), where participants stand barefoot with arms at their sides for two 30-second trials each
Sit-to-stand | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The sit-to-stand test requires participants to rise as quickly as possible from a seated position with 90º knee flexion and arms crossed
Sit-to-stand | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The sit-to-stand test requires participants to rise as quickly as possible from a seated position with 90º knee flexion and arms crossed
Timed Up-and-Go test | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  In the Timed Up-and-Go test, participants move from sitting to standing, walk 3 meters, turn, return, and sit
Timed Up-and-Go test | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  In the Timed Up-and-Go test, participants move from sitting to standing, walk 3 meters, turn, return, and sit
Delayed onset muscle soreness | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  To measure delayed onset muscle soreness (DOMS), a 10-point visual analogue scale shall be used, where 1 = no pain and 10 = intolerable pain
Delayed onset muscle soreness | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  To measure delayed onset muscle soreness (DOMS), a 10-point visual analogue scale shall be used, where 1 = no pain and 10 = intolerable pain
Delayed onset muscle soreness | Post-intervention (24 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  To measure delayed onset muscle soreness (DOMS), a 10-point visual analogue scale shall be used, where 1 = no pain and 10 = intolerable pain
Delayed onset muscle soreness | Post-intervention (48 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  To measure delayed onset muscle soreness (DOMS), a 10-point visual analogue scale shall be used, where 1 = no pain and 10 = intolerable pain
Delayed onset muscle soreness | Post-intervention (72 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  To measure delayed onset muscle soreness (DOMS), a 10-point visual analogue scale shall be used, where 1 = no pain and 10 = intolerable pain
Subjective Perception of Effort (RPE) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Participants will be instructed and familiarized with the use of the Borg Rating of Perceived Exertion scale during the familiarization phase. Subjective perception of effort will be assessed before, during (after each exercise within the session), and after the training session using the Borg Rating of Perceived Exertion Scale (6-20 points). On this scale, 6 indicates "no exertion at all" and 20 indicates "maximal exertion". Higher scores represent greater perceived effort.
Subjective Perception of Effort | Post-intervention (24 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Participants will be instructed and familiarized with the use of the RPE scale during the familiarization phase. RPE will be assessed before, during (after each exercise within the session), and after the training session using the Borg 6-20 RPE scale
Subjective Perception of Effort | Post-intervention (48 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Participants will be instructed and familiarized with the use of the RPE scale during the familiarization phase. RPE will be assessed before, during (after each exercise within the session), and after the training session using the Borg 6-20 RPE scale
Subjective Perception of Effort | Post-intervention (72 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Participants will be instructed and familiarized with the use of the RPE scale during the familiarization phase. RPE will be assessed before, during (after each exercise within the session), and after the training session using the Borg 6-20 RPE scale
Fatigue Visual Analog Scale (VAS-F) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The VAS-F will be used to measure fatigue. This scale, is subdivided into two subscales: fatigue and energy. The VAS-F features a 100 mm long horizontal line, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line corresponding to their perception of the severity of fatigue between these two endpoints.
Visual Analogue Scale for Fatigue (VAS-F) | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The VAS-F will be used to measure fatigue. This scale, is subdivided into two subscales: fatigue and energy. The VAS-F features a 100 mm long horizontal line, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line corresponding to their perception of the severity of fatigue between these two endpoints.
Fatigue Visual Analog Scale (VAS-F) | Post-intervention (24 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The VAS-F will be used to measure fatigue. This scale, is subdivided into two subscales: fatigue and energy. The VAS-F features a 100 mm long horizontal line, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line corresponding to their perception of the severity of fatigue between these two endpoints.
Fatigue Visual Analog Scale (VAS-F) | Post-intervention (48 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The VAS-F will be used to measure fatigue. This scale, is subdivided into two subscales: fatigue and energy. The VAS-F features a 100 mm long horizontal line, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line corresponding to their perception of the severity of fatigue between these two endpoints.
Fatigue Visual Analog Scale (VAS-F) | Post-intervention (72 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  The VAS-F will be used to measure fatigue. This scale, is subdivided into two subscales: fatigue and energy. The VAS-F features a 100 mm long horizontal line, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line corresponding to their perception of the severity of fatigue between these two endpoints.
Body Weight | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Body weight will be measured using a calibrated digital scale. The participant will be barefoot and wearing light clothing.
  Unit of Measure: Kilograms (kg)
Physical Activity Level assessed by the International Physical Activity Questionnaire (IPAQ) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Physical activity will be assessed using the IPAQ (short form), adapted for people with multiple sclerosis. The questionnaire captures frequency and duration of physical activity in walking, moderate, and vigorous domains over the last 7 days. MET values will be adjusted for the functional limitations commonly present in this population. Unit of Measure: MET-minutes per week
Adherence to the Mediterranean Diet assessed by MEDAS | Baseline (pre-intervention)
  Adherence to the Mediterranean Diet will be assessed using the MEDAS (Mediterranean Diet Adherence Screener), a validated 14-item questionnaire designed to evaluate dietary patterns. The questionnaire measures adherence based on the consumption of key food groups associated with the Mediterranean diet. Unit of Measure: Score on the MEDAS questionnaire (range: 0-14; higher scores indicate greater adherence)
Adherence to the Mediterranean Diet assessed by MEDAS | Post-intervention (48 hours after the last session)
  Adherence to the Mediterranean Diet will be assessed using the MEDAS (Mediterranean Diet Adherence Screener), a validated 14-item questionnaire designed to evaluate dietary patterns. The questionnaire measures adherence based on the consumption of key food groups associated with the Mediterranean diet. Unit of Measure: Score on the MEDAS questionnaire (range: 0-14; higher scores indicate greater adherence)
The Kurtzke Disability Scale | Baseline (pre-intervention).
  The Kurtzke Disability Scale (EDSS) is divided into 8 functional systems (FS); four primary: pyramidal function, cerebellar function, sensory function, and brainstem function; and four secondary: sphincters, vision, mental, and others. For each FS, a severity score is provided, ranging from 0 to 6 or 7. The overall score of the scale is measured on a 20-item scale (from 0 to 10 points, increasing in half-point increments). Up to 3.5, the score obtained in each FS and the number of affected FS automatically determine the EDSS score. From 4 to 7, the definition of each level is also given by the ability to walk (ability to walk without stopping, need for assistance) Time Frame: Before the first session of the intervention program
The Kurtzke Disability Scale | Post-intervention (48 hours after the last session).
  The Kurtzke Disability Scale (EDSS) is divided into 8 functional systems (FS); four primary: pyramidal function, cerebellar function, sensory function, and brainstem function; and four secondary: sphincters, vision, mental, and others. For each FS, a severity score is provided, ranging from 0 to 6 or 7. The overall score of the scale is measured on a 20-item scale (from 0 to 10 points, increasing in half-point increments). Up to 3.5, the score obtained in each FS and the number of affected FS automatically determine the EDSS score. From 4 to 7, the definition of each level is also given by the ability to walk (ability to walk without stopping, need for assistance) Time Frame: Before the first session of the intervention program
Subjective Sleep Quality Questionnaire | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnaire [73]. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (woke up too early [1] - did not wake up early [3]), e) ease of waking up (very difficult [1] - very easy [5]), f) feeling of rest (did not rest at all [1] - fully rested [3]), and g) sufficient sleep (no, definitely too little [1] - yes, definitely enough [5]).
Subjective Sleep Quality Questionnaire | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnaire [73]. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (woke up too early [1] - did not wake up early [3]), e) ease of waking up (very difficult [1] - very easy [5]), f) feeling of rest (did not rest at all [1] - fully rested [3]), and g) sufficient sleep (no, definitely too little [1] - yes, definitely enough [5]).
Subjective Sleep Quality Questionnaire | Post-intervention (24 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnaire [73]. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (woke up too early [1] - did not wake up early [3]), e) ease of waking up (very difficult [1] - very easy [5]), f) feeling of rest (did not rest at all [1] - fully rested [3]), and g) sufficient sleep (no, definitely too little [1] - yes, definitely enough [5]).
  Time Frame: Before the first session of the intervention program
Subjective Sleep Quality Questionnaire | Post-intervention (48 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnaire [73]. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (woke up too early [1] - did not wake up early [3]), e) ease of waking up (very difficult [1] - very easy [5]), f) feeling of rest (did not rest at all [1] - fully rested [3]), and g) sufficient sleep (no, definitely too little [1] - yes, definitely enough [5]).
  Time Frame: Before the first session of the intervention program
Subjective Sleep Quality Questionnaire | Post-intervention (72 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnaire [73]. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (woke up too early [1] - did not wake up early [3]), e) ease of waking up (very difficult [1] - very easy [5]), f) feeling of rest (did not rest at all [1] - fully rested [3]), and g) sufficient sleep (no, definitely too little [1] - yes, definitely enough [5]).
  Time Frame: Before the first session of the intervention program
Sleep Quality Measured by Actigraph | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Sleep quality based on actigraphy will be evaluated using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK) [74]. This device uses a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower sensitivity threshold for actigraphy will be set at 80 counts/epoch. Data analysis will begin at the start of the nighttime rest period (bedtime) and conclude at the start of daytime activity (wake-up time)
Sleep Quality Measured by Actigraph | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Sleep quality based on actigraphy will be evaluated using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK) [74]. This device uses a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower sensitivity threshold for actigraphy will be set at 80 counts/epoch. Data analysis will begin at the start of the nighttime rest period (bedtime) and conclude at the start of daytime activity (wake-up time)
Sleep Quality Measured by Actigraph | Post-intervention (24 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Sleep quality based on actigraphy will be evaluated using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK) [74]. This device uses a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower sensitivity threshold for actigraphy will be set at 80 counts/epoch. Data analysis will begin at the start of the nighttime rest period (bedtime) and conclude at the start of daytime activity (wake-up time)
Sleep Quality Measured by Actigraph | Post-intervention (48 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Sleep quality based on actigraphy will be evaluated using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK) [74]. This device uses a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower sensitivity threshold for actigraphy will be set at 80 counts/epoch. Data analysis will begin at the start of the nighttime rest period (bedtime) and conclude at the start of daytime activity (wake-up time)
Sleep Quality Measured by Actigraph | Post-intervention (72 hours after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Sleep quality based on actigraphy will be evaluated using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK) [74]. This device uses a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower sensitivity threshold for actigraphy will be set at 80 counts/epoch. Data analysis will begin at the start of the nighttime rest period (bedtime) and conclude at the start of daytime activity (wake-up time)
Progesterone (PG) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Serum progesterone levels will be measured to confirm luteal phase and ovulatory patterns. Unit of measure: ng/mL
Luteinizing Hormone (LH) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  LH will be measured to detect the ovulatory surge and determine phase timing. Unit of measure: mIU/mL
Follicle-Stimulating Hormone (FSH) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  FSH levels will be assessed to evaluate ovarian function. Unit of measure: mIU/mL
Estradiol (E2) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Serum estradiol will be analyzed to confirm hormonal variation across the menstrual cycle. Unit of measure: pg/mL
Testosterone (T) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Serum testosterone will be measured to examine androgen levels. Unit of measure: ng/dL
Interleukin-6 (IL-6) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Serum IL-6 will be measured to evaluate systemic inflammation. Unit of measure: pg/mL
Interleukin-6 (IL-6) | Post-intervention (30 min after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Serum IL-6 will be measured to evaluate systemic inflammation. Unit of measure: pg/mL
Tumor Necrosis Factor-alpha (TNF-α) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  TNF-α levels will be assessed as an indicator of inflammatory status. Unit of measure: pg/mL
Tumor Necrosis Factor-alpha (TNF-α) | Post-intervention (30 min after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  TNF-α levels will be assessed as an indicator of inflammatory status. Unit of measure: pg/mL
Interleukin-10 (IL-10) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  IL-10 will be measured to evaluate anti-inflammatory responses. Unit of measure: pg/mL
Interleukin-10 (IL-10) | Post-intervention (30 min after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  IL-10 will be measured to evaluate anti-inflammatory responses. Unit of measure: pg/mL
Transforming Growth Factor Beta 1 (TGF-β1) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  TGF-β1 levels will be analyzed as part of the immunomodulatory and regulatory response profile.
  Unit of measure: ng/mL
Transforming Growth Factor Beta 1 (TGF-β1) | Post-intervention (30 min after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  TGF-β1 levels will be analyzed as part of the immunomodulatory and regulatory response profile. Unit of measure: ng/mL
Intrinsic muscle characteristics: Stiffness (S) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Stiffness assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia). Definition: dynamic stiffness (N/m) characterizes the resistance of biological soft tissues to a force of deformation
Intrinsic muscle characteristics: Stiffness (S) | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Stiffness assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia). Definition: dynamic stiffness (N/m) characterizes the resistance of biological soft tissues to a force of deformation
Intrinsic muscle characteristics: Elasticity (D) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Elasticity assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia). Definition elasticity: logarithmic decrement (arb) characterizes the dampening of tissue oscillation.
Intrinsic muscle characteristics: Elasticity (D) | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Elasticity assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia). Definition elasticity: logarithmic decrement (arb) characterizes the dampening of tissue oscillation
Intrinsic muscle characteristics: Relaxation (R) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Relaxation assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia). Definition relaxation: Mechanical stress relaxation time (ms) characterizes tissue´s recovery time from displacement.
Intrinsic muscle characteristics: Relaxation (R) | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Relaxation assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia). Definition relaxation: Mechanical stress relaxation time (ms) characterizes tissue´s recovery time from displacement.
Intrinsic muscle characteristics: Creep (C) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Creep assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia). Definition creep: ratio of relaxation and deformation time (arb) characterizes creep, the gradual elongation of tissue over time when placed under constant tensile stress.
Intrinsic muscle characteristics: Creep (C) | Post-intervention (immediately after) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Creep assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia). Definition creep: ratio of relaxation and deformation time (arb) characterizes creep, the gradual elongation of tissue over time when placed under constant tensile stress.
Height | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Height will be measured using a wall-mounted stadiometer with the participant barefoot and standing upright.
  Unit of Measure: Meters (m)
Body Mass Index (BMI) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  BMI will be calculated as weight in kilograms divided by the square of height in meters (kg/m²). Body weight and height will be assessed using a calibrated digital scale and stadiometer, respectively.
Physical Activity Level assessed by Triaxial Accelerometer | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Objective physical activity will be measured using a triaxial accelerometer, which captures movement in three planes (vertical, lateral, and anterior-posterior). Variables include time spent in light, moderate, and vigorous physical activity, as well as step count. This tool enables detailed quantification of low-intensity movements common in individuals with MS. Unit of Measure: Minutes per day in activity categories; steps per day
Nutrient Intake assessed by 3-Day Food Diary | Baseline (pre-intervention)
  Dietary intake will be assessed using a 3-day food diary, including two weekdays and one weekend day. Participants will record all food and beverages consumed, and a registered dietitian will analyze macronutrient and micronutrient intake using nutrition software. Unit of Measure: Daily intake in grams (carbohydrates, proteins, fats) and milligrams/micrograms (vitamins, minerals), as appropriate
Nutrient Intake assessed by 3-Day Food Diary | Post-intervention (48 hours after the last session)
  Dietary intake will be assessed using a 3-day food diary, including two weekdays and one weekend day. Participants will record all food and beverages consumed, and a registered dietitian will analyze macronutrient and micronutrient intake using nutrition software. Unit of Measure: Daily intake in grams (carbohydrates, proteins, fats) and milligrams/micrograms (vitamins, minerals), as appropriate
Lean Mass (%) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Lean mass will be evaluated using BIA and DXA, both for the entire body and segmentally (arms, legs, trunk). Unit of Measure: %
Lean Mass (kg) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Lean mass will be evaluated using BIA and DXA, both for the entire body and segmentally (arms, legs, trunk). Unit of Measure: kilograms
Bone Mineral Content (BMC) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Bone Mineral Content will be measured using DXA, both globally and at specific body segments (e.g., spine, hips, limbs). BMC indicates the total mineral content in bones and is essential for assessing bone health in MS. Unit of Measure: Grams (g)
Bone Mineral Density (BMD) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Bone Mineral Density will be assessed with DXA, capturing whole-body and segmental (lumbar spine, femoral neck, etc.) density in g/cm². BMD reflects bone strength and fracture risk.
  Unit of Measure: g/cm²
Body Water | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Total body water will be measured using BIA, evaluating both intracellular and extracellular compartments. Segmental analysis (e.g., limbs and trunk) will also be included to reflect fluid distribution patterns. Unit of Measure: Liters (L)
Phase Angle | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Phase angle will be assessed with BIA for both total and segmental body regions. It reflects cellular health and membrane integrity, and is an important marker of nutritional and physiological status in MS patients. Unit of Measure: Degrees (°)
Heart rate variability | Post-intervention (first night) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  HRV measurements will be taken using a Polar H10 heart rate sensor (Kempele, Finland), which participants will be instructed to wear when going to bed. The sensor will record heartbeats during sleep, and the data will be analyzed using Kubios HRV software (version 3.0). The Poincaré plot and time and frequency domains will be analyzed.
Heart rate variability | Post-intervention (24 hours after, i.e., the second night) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  HRV measurements will be taken using a Polar H10 heart rate sensor (Kempele, Finland), which participants will be instructed to wear when going to bed. The sensor will record heartbeats during sleep, and the data will be analyzed using Kubios HRV software (version 3.0). The Poincaré plot and time and frequency domains will be analyzed.
Heart rate variability | Post-intervention (48 hours after, i.e., the third night) in each menstrual phase: early follicular (Days 2-5), late follicular (Days -2 to 0, LH peak), and mid-luteal (Days 6-9 after LH peak).
  HRV measurements will be taken using a Polar H10 heart rate sensor (Kempele, Finland), which participants will be instructed to wear when going to bed. The sensor will record heartbeats during sleep, and the data will be analyzed using Kubios HRV software (version 3.0). The Poincaré plot and time and frequency domains will be analyzed.
Heart rate variability | Post-intervention (72 hours after, i.e., the fourth night) in each menstrual phase: early follicular (Days 2-5), late follicular (Days -2 to 0, LH peak), and mid-luteal (Days 6-9 after LH peak).
  HRV measurements will be taken using a Polar H10 heart rate sensor (Kempele, Finland), which participants will be instructed to wear when going to bed. The sensor will record heartbeats during sleep, and the data will be analyzed using Kubios HRV software (version 3.0). The Poincaré plot and time and frequency domains will be analyzed.
Fat Mass (kg) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Fat mass will be measured using bioelectrical impedance analysis (BIA) and dual-energy X-ray absorptiometry (DXA). Both whole-body and segmental (arms, legs, trunk) fat mass will be assessed. Unit of Measure: Kilograms
Fat Mass (%) | Pre-intervention (immediately before) in each menstrual phase: Early follicular (Days 2-5), Late follicular (Days -2 to 0, LH peak), and Mid-luteal (Days 6-9 after LH peak).
  Fat mass will be measured using bioelectrical impedance analysis (BIA) and dual-energy X-ray absorptiometry (DXA). Both whole-body and segmental (arms, legs, trunk) fat mass will be assessed. Unit of Measure: %

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen de la Arrixaca, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided